CLINICAL TRIAL: NCT05247359
Title: Neuromuscular Deficits in Jump-Landing Technique in Young Basketball: a Cross-sectional Observational Study
Brief Title: Neuromuscular Deficits in Jump-Landing Technique in Young Basketball
Acronym: ALFUSABA
Status: Completed | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Associate Professor, University Rovira i Virgili
Other Study IDs: CEIPSA-2021-PR-0009
Record Dates: First submitted 2022-01-28; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Sport Injury; Motor Skills Disorders; Biomechanical Lesions
Keywords: Basketball; Physical Therapy; Youth athletes; Movement
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Basketball is a team sport that requires specific motor skills to develop different technical-tactical actions. Within the specific movements, landings after a jump are very common and require optimal technical performance, good stability and symmetry. Alterations in these components have been linked to an increased risk of injury. The objective of the present study is to identify functional alterations in the jump / landing technique that basketball players present.

Cross-sectional study carried out from Septembre to Juny. The participants were basketball players aged 12 to 14 years. The main variables were: ankle stability, dynamic knee valgus, central stability, symmetry of the lower extremities. The tests used were: Abalakov Test, Single Hop Test for distance, Single-leg vertical countermovement jump test, Cross Over Hop test, One Leg Balance Test.

DETAILED DESCRIPTION:
Basketball is a team sport that requires specific motor skills to develop different technical-tactical actions. Within the specific movements, landings after a jump are very common and require optimal technical performance, good stability and symmetry. Alterations in these components have been linked to an increased risk of injury. The objective of the present study is to identify functional alterations in the jump / landing technique that basketball players present. A cross-sectional study carried out from Septembre to Juny. The participants were basketball players aged 12 to 14 years. The main variables were: ankle stability, dynamic knee valgus, central stability, symmetry of the lower extremities. The tests used were: Abalakov Test, Single Hop Test for distance, Single-leg vertical countermovement jump test, Cross Over Hop test, One Leg Balance Test.

ELIGIBILITY:
Inclusion Criteria:

* Age from 12 years to 14 years at testing (both included).
* To be actively competing during the study.
* Voluntarily sign the informed consent form.
* Not meet the exclusion criteria.

Exclusion Criteria:

* Presented any injury (overuse or acute) at the time of testing.
* Psychological or psychiatric diseases diagnosed.
* Oncological diseases diagnosed.
* Did not attend on the day of the assessment.

Ages: 12 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: The participants were recruited through the Catalan Basketball Federation, and the study was carried out in the sports facilities of each club.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Ankle stability | 1 year
  The ability of the player to maintain the monopodal position throughout the test and at the same time perform the jumps continuously without compensating with small jumps to stabilize was evaluated with the Cross Over Hop test and Single Hop Test for distance. It was recorded with a frontal and lateral filming device. The results were subsequently analyzed.
Dynamic lower extremity valgus | 1 year
  It was evaluated with the Abalakov Test and the Single Hop test for distance. For this purpose, two filming devices were placed, one frontal and one lateral. For the detection of dynamic valgus at landing, the angle formed between the femur and the tibia was looked at. The results were subsequently analyzed with the recording obtained.
Dynamic postural control | 1 year
  The Abalakov Test, Single Hop Test for distance and the Single-leg vertical countermovement jump test were used to observe the trunk alignment during the jump taking the hip and shoulder girdle as reference. For this purpose, two filming devices were placed in frontal and lateral positions. The results were subsequently analyzed with the recording obtained.
Symmetry | 1 year
  From the distance obtained in the Single Hop for distance Test, the Symmetry Index was calculated through the formula: (Distance dominant limb/Distance non-dominant limb)*100.

SECONDARY OUTCOMES:
Age | 1 year
  Years
Gender | 1 year
  Female or male
Weight | 1 year
  A scale accurate to +100 kg was used. The weight of the subject, barefoot and in training clothes, was recorded in Kg.
Height | 1 year
  A centimeter tape placed on the wall was used. The height was recorded in meters. For this purpose, the player stood barefoot and with the back of the heels, shoulders and head in contact with the wall. Maintaining an upright position, the entire sole of the foot in contact with the floor, and looking straight ahead.
Wingspan | 1 year
  A centimeter tape attached to the wall in a horizontal position at the height of each player's shoulders was used. The subject was positioned barefoot and with the back of the heels, shoulders and head in contact with the wall. The arms were placed in 90o abduction, with slight external rotation, thumbs up and hand open. Always maintaining an upright position, the entire sole of the foot in contact with the floor, and the gaze facing forward. The result was recorded in meters.
Speed | 1 year
  It was evaluated with the 30m sprint test and a stopwatch was used to record the time (in seconds) it took the player to run 30 meters in a straight line at the fastest possible speed. Two attempts were made and the best time was recorded. For the test to be valid, the player did not have to start the race before the starting signal, nor had to have the foot advanced beyond the starting line.
Agility | 1 year
  The Lane Agility Test drill was used. The time (in seconds) it took the player to traverse the rectangle formed by the 4 cones, first in one direction and then in the other, was timed.
Power | 1 year
  It was evaluated with the Single-leg vertical countermovement jump test and the Chronojump force platform. Lower extremity power was recorded in watts.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Adillón, MsC, Principal Investigator — University Rovira i Virgili
Locations (1):
- Federación Catalana de Baloncesto, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baltaci G, Yilmaz G, Atay AO. The outcomes of anterior cruciate ligament reconstructed and rehabilitated knees versus healthy knees: a functional comparison. Acta Orthop Traumatol Turc. 2012;46(3):186-95. doi: 10.3944/aott.2012.2366. PMID 22659635
- [Background] Lee DW, Yang SJ, Cho SI, Lee JH, Kim JG. Single-leg vertical jump test as a functional test after anterior cruciate ligament reconstruction. Knee. 2018 Dec;25(6):1016-1026. doi: 10.1016/j.knee.2018.07.014. Epub 2018 Aug 14. PMID 30115591
- [Background] Fernandez-Santos JR, Ruiz JR, Cohen DD, Gonzalez-Montesinos JL, Castro-Pinero J. Reliability and Validity of Tests to Assess Lower-Body Muscular Power in Children. J Strength Cond Res. 2015 Aug;29(8):2277-85. doi: 10.1519/JSC.0000000000000864. PMID 25647647
- [Background] Read PJ, Oliver JL, de Ste Croix MB, Myer GD, Lloyd RS. Reliability of the Tuck Jump Injury Risk Screening Assessment in Elite Male Youth Soccer Players. J Strength Cond Res. 2016 Jun;30(6):1510-6. doi: 10.1519/JSC.0000000000001260. PMID 26562715
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Troester JC, Jasmin JG, Duffield R. Reliability of Single-Leg Balance and Landing Tests in Rugby Union; Prospect of Using Postural Control to Monitor Fatigue. J Sports Sci Med. 2018 May 14;17(2):174-180. eCollection 2018 Jun. PMID 29769817
- [Background] Jonsson E, Seiger A, Hirschfeld H. One-leg stance in healthy young and elderly adults: a measure of postural steadiness? Clin Biomech (Bristol). 2004 Aug;19(7):688-94. doi: 10.1016/j.clinbiomech.2004.04.002. PMID 15288454
- [Background] Michikawa T, Nishiwaki Y, Takebayashi T, Toyama Y. One-leg standing test for elderly populations. J Orthop Sci. 2009 Sep;14(5):675-85. doi: 10.1007/s00776-009-1371-6. Epub 2009 Oct 3. PMID 19802686
- [Background] Lockie RG, Beljic A, Ducheny SC, Kammerer JD, Dawes JJ. Relationships between Playing Time and Selected NBA Combine Test Performance in Division I Mid-Major Basketball Players. Int J Exerc Sci. 2020 May 1;13(4):583-596. doi: 10.70252/XZEP5232. eCollection 2020. PMID 32509125
- [Background] Stojanovic E, Aksovic N, Stojiljkovic N, Stankovic R, Scanlan AT, Milanovic Z. Reliability, Usefulness, and Factorial Validity of Change-of-direction Speed Tests in Adolescent Basketball Players. J Strength Cond Res. 2019 Nov;33(11):3162-3173. doi: 10.1519/JSC.0000000000002666. PMID 29927890
- [Background] Fort-Vanmeerhaeghe A, Tutusaus L, Ruiz P, Massó i Ortigosa N. Efectos de un entrenamiento propioceptivo sobre la extremidad inferior en jóvenes deportistas jugadores de voleibol. Apunts. Medicina de l'Esport. 2008;43(157):5-13.
- [Result] Harmer PA. Basketball injuries. Med Sport Sci. 2005;49:31-61. doi: 10.1159/000085341. PMID 16247261
- [Result] Fort-Vanmeerhaeghe A, Romero Rodriguez D. Análisis de los factores de riesgo neuromusculares de las lesiones deportivas. Apunts Med l Esport. 2013;48(179):109- 120.
- [Result] Schelling X, Torres-Ronda L. An integrative approach to stenght and neuromuscular power training for basketball. Strenghth & Conditioning Journal. 2016;38(3):72-80.
- [Result] Policastro F, Accardo A, Marcovich R, Pelamatti G, Zoia S. Relation between Motor and Cognitive Skills in Italian Basketball Players Aged between 7 and 10 Years Old. Sports (Basel). 2018 Aug 14;6(3):80. doi: 10.3390/sports6030080. PMID 30110977
- [Result] Stelee J, Sheppard J. Landing mechanics in injury prevention and performance rehabilitation. In: Joyce D, Lewindon D. Sports Injury Prevention and Rehabilitation: integrating medicine and science for performance solutions. London: Taylor & Francis Group; 2016:121-138.
- [Result] Struzik A, Juras G, Pietraszewski B, Rokita A. Effect of drop jump technique on the reactive strength index. J Hum Kinet. 2016 Sep 10;52:157-164. doi: 10.1515/hukin-2016-0003. eCollection 2016 Sep 1. PMID 28149403
- [Result] Romanchuk NJ, Smale KB, Del Bel MJ, Benoit DL. Divergence analysis of failed and successful unanticipated single-leg landings reveals the importance of the flight phase and upper body biomechanics. J Biomech. 2020 Aug 26;109:109879. doi: 10.1016/j.jbiomech.2020.109879. Epub 2020 Jun 13. PMID 32807323
- [Result] Sugiyama T, Kameda M, Kageyama M, Kiba K, Kanehisa H, Maeda A. Asymmetry between the Dominant and Non-Dominant Legs in the Kinematics of the Lower Extremities during a Running Single Leg Jump in Collegiate Basketball Players. J Sports Sci Med. 2014 Dec 1;13(4):951-7. eCollection 2014 Dec. PMID 25435790
- [Result] Fort-Vanmeerhaeghe A, Bishop C, Busca B, Aguilera-Castells J, Vicens-Bordas J, Gonzalo-Skok O. Inter-limb asymmetries are associated with decrements in physical performance in youth elite team sports athletes. PLoS One. 2020 Mar 3;15(3):e0229440. doi: 10.1371/journal.pone.0229440. eCollection 2020. PMID 32126107
- [Result] Fort-Vanmeerhaeghe A, Montalvo AM, Lloyd RS, Read P, Myer GD. Intra- and Inter-Rater Reliability of the Modified Tuck Jump Assessment. J Sports Sci Med. 2017 Mar 1;16(1):117-124. eCollection 2017 Mar. PMID 28344460
- [Result] Caffrey E, Docherty CL, Schrader J, Klossner J. The ability of 4 single-limb hopping tests to detect functional performance deficits in individuals with functional ankle instability. J Orthop Sports Phys Ther. 2009 Nov;39(11):799-806. doi: 10.2519/jospt.2009.3042. PMID 19881005
- [Result] Gillen ZM, Shoemaker ME, McKay BD, Bohannon NA, Gibson SM, Cramer JT. Influences of the Stretch-Shortening Cycle and Arm Swing on Vertical Jump Performance in Children and Adolescents. J Strength Cond Res. 2022 May 1;36(5):1245-1256. doi: 10.1519/JSC.0000000000003647. Epub 2020 May 28. PMID 32483060
- [Result] Sasaki S, Tsuda E, Yamamoto Y, Maeda S, Kimura Y, Fujita Y, Ishibashi Y. Core-Muscle Training and Neuromuscular Control of the Lower Limb and Trunk. J Athl Train. 2019 Sep;54(9):959-969. doi: 10.4085/1062-6050-113-17. Epub 2019 Aug 6. PMID 31386583
- [Result] Mackala K, Stodolka J, Siemienski A, Coh M. Biomechanical analysis of squat jump and countermovement jump from varying starting positions. J Strength Cond Res. 2013 Oct;27(10):2650-61. doi: 10.1519/JSC.0b013e31828909ec. PMID 23552341
- [Result] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287
- [Result] Agel J, Olson DE, Dick R, Arendt EA, Marshall SW, Sikka RS. Descriptive epidemiology of collegiate women's basketball injuries: National Collegiate Athletic Association Injury Surveillance System, 1988-1989 through 2003-2004. J Athl Train. 2007 Apr-Jun;42(2):202-10. PMID 17710168
- [Result] Ford KR, Myer GD, Hewett TE. Valgus knee motion during landing in high school female and male basketball players. Med Sci Sports Exerc. 2003 Oct;35(10):1745-50. doi: 10.1249/01.MSS.0000089346.85744.D9. PMID 14523314
- [Result] Randazzo C, Nelson NG, McKenzie LB. Basketball-related injuries in school-aged children and adolescents in 1997-2007. Pediatrics. 2010 Oct;126(4):727-33. doi: 10.1542/peds.2009-2497. Epub 2010 Sep 13. PMID 20837592